CLINICAL TRIAL: NCT06260839
Title: Evaluation of the Effect of Percutaneous Minimally Invasive Technique Assisted by Magnetic Resonance Neurography in the Treatment of Gluteal Muscle Contracture
Brief Title: the Effect of Minimally Invasive Technique Assisted by Magnetic Resonance Neurography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Xiang (Other)
Responsible Party: Sponsor-Investigator, He Xiang, The First Affiliated Hospital of Air Force Medicial University, The First Affiliated Hospital of Air Force Medicial University
Organization: The First Affiliated Hospital of Air Force Medicial University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20232442-F-1
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Orthopedic Surgery
Keywords: gluteal muscle contracture; Minimally invasive release surgery; Magnetic resonance neurography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRN guided minimally invasive surgery group (Experimental): The intervention measures of the experimental group were to analyze the relationship between the shape of the contracture band, the distance between the sciatic nerve and the contracture band, and the external rotation angle according to the preoperative MRN manifestations of the patients, and to design the individualized surgical approach according to the imaging manifestations and perform MRN-assisted minimally invasive release.
  Interventions: Procedure: magnetic resonance neurography
- Minimally invasive surgery group (Active Comparator): In the control group, preoperative magnetic resonance imaging was only used to assist in the diagnosis and evaluation of gluteal muscle contracture, and the results of magnetic resonance imaging were not used to assist in the design of surgical approach. In the control group, non-MRN-assisted minimally invasive release was performed
  Interventions: Procedure: no magnetic resonance neurography

INTERVENTIONS:
Procedure: magnetic resonance neurography — preoperative magnetic resonance neurography and assisted design of surgical approach
  Arms: MRN guided minimally invasive surgery group
Procedure: no magnetic resonance neurography — Preoperative magnetic resonance neurography was not performed, and general minimally invasive surgery was performed
  Arms: Minimally invasive surgery group

SUMMARY:
The goal of this clinical trial is to to compare the therapeutic effect of minimally invasive surgery guided by magnetic resonance neurography(MRN) compared with non-magnetic resonance assisted minimally invasive surgery in patients with moderate to severe gluteal muscle contracture(GMC). The main question it aims to answer are: magnetic resonance neurography can better help optimize the surgical path of minimally invasive surgery in the treatment of gluteal muscle contracture.

Participants will underwent preoperative magnetic resonance examination according to different groups, and then the experimental group designed individualized surgical approach and MRN-assisted minimally invasive release according to the imaging findings. In the control group, preoperative magnetic resonance examination was only used to assist in the diagnosis and evaluation of gluteal muscle contracture, and the magnetic resonance results were not used to assist in the design of surgical approach. In the control group, non-MRN-assisted minimally invasive release was performed. The researchers will compare the intraoperative surgery-related indicators and postoperative hip function scores and complications of patients in different groups to see if magnetic resonance-assisted surgery has a better postoperative effect.

DETAILED DESCRIPTION:
According to the different surgical intervention methods, the cases finally included in the study were divided into minimally invasive surgery group and MRN-guided minimally invasive surgery group according to the randomization method. It is expected that the number of cases finally included in the study in both groups will be 22 cases.

Firstly, the age and sex of the two groups of patients included in the study were recorded respectively, and the moderate and severe classification was carried out according to the Zhao 's classification system. The experimental group and the control group were examined by pelvic X-ray, magnetic resonance and ultrasound before operation. After improving the relevant preoperative examination and excluding surgical contraindications, the intervention measures of the experimental group were to analyze the relationship between the shape of the contracture zone, the distance between the sciatic nerve and the contracture zone, and the external rotation angle according to the preoperative MRN manifestations of the patients, and to design the individualized surgical approach according to the imaging manifestations. MRN-assisted minimally invasive release ; in the control group, preoperative magnetic resonance imaging was only used to assist in the diagnosis and evaluation of gluteal muscle contracture, and the results of magnetic resonance imaging were not used to assist in the design of surgical approach. In the control group, non-MRN-assisted minimally invasive release was performed. For patients, they all underwent magnetic resonance imaging before surgery, and all underwent minimally invasive surgery. However, the design process of the specific surgical approach is not clear, so it is a single-blind design for patients. All the operations were completed by two senior doctors of our research group. The data of postoperative follow-up were recorded, and the conclusion was drawn by statistical analysis.

Intraoperative research indicators include : incision length, operation duration, intraoperative blood loss, first time to get out of bed, pain score, etc.

Postoperative follow-up study indicators included : subjective and objective functional rating scales ( hip flexion and adduction activity, leg squat, cross-leg test, Ober sign, pain in activity, claudication in walking ), patient appearance satisfaction, complications ( wound infection, fat liquefaction, neurovascular injury, incision hematoma formation, etc. ).

ELIGIBILITY:
Inclusion Criteria：

（1). Meet the clinical and imaging diagnostic criteria of GMC ; (2).According to Zhao 's classification system, patients with moderate to severe GMC diagnosed by medical history, symptoms and physical examination ; (3).Conservative treatment is ineffective for at least 6 months, and daily life is significantly affected ; (4).willing to be hospitalized and receive minimally invasive surgery ; (5). Can cooperate to complete the follow-up ; (6).Patients or immediate family members signed informed consent ; (7). Age 18-65 years old

Exclusion Criteria:

1. . There is clinical or imaging evidence that there is or may be spinal or lower extremity neurological disease ;
2. . There is evidence of hip dysplasia or subluxation ;
3. .after evaluation of intolerance to surgical anesthesia ;
4. .coagulant dysfunction ;
5. . unable to complete the follow-up for various reasons ;
6. . Patients can not complete the scale assessment for other reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hip joint outcome score(HOS) scale | one week after operation
  The hip joint outcome score ( HOS ) was divided into two parts : the activities-of-daily-living ( HOS-ADL ) and sports subscales( HOS-SS ).The lowest score of the scale was 0, and the highest score was 100. The higher the final score, the higher the level of daily life and motor function of hip joint.
Objective hip function scoring scale | one week after operation
  The objective hip function scoring scale is a scale used to objectively evaluate the function of hip joint. The hip joint function of patients is evaluated by doctors and scored one by one according to the items. The lowest score of the scale was 0, and the highest score was 100. The higher the final score, the better the hip joint function.

SECONDARY OUTCOMES:
Hip joint function of patients | One day before surgery and three days after surgery
  The patient 's hip function is mainly evaluated by the physician during physical examination. The main indicators include hip flexion and adduction activity, and leg squat, cross-legged test, Ober sign, activity with or without pain, walking with or without claudication.
Imaging data of patients with gluteal muscle contracture | One day before surgery and three days after surgery
  The imaging data of the patients included the presence or absence of gluteus maximus atrophy, the cumulative range of the contracture zone, the characteristics of the course, and the presence or absence of connection with the iliotibial tract ; the distance between the contracture belt and the sciatic nerve ; external rotation angle of femur.
Record the duration of the patient 's surgery | During surgery
  Through the operation record, nursing record and the actual situation of the operation, the operation duration of the patients was recorded. The longer the operation duration, the greater the operation risk.
The record of the length of the surgical incision of the patient | During surgery
  Through the patient 's surgical records and intraoperative actual situation, record the patient 's intraoperative incision length. The greater the length of the incision, the greater the risk of surgery.
Measurement of intraoperative blood loss | During surgery
  The patient 's intraoperative blood loss was recorded through the patient 's anesthesia records, nursing records, and actual intraoperative conditions. The higher the amount of bleeding, the greater the risk of surgery.
The first ambulation time after operation | The second day after surgery
  The time when the patient can get out of bed for the first time after surgery, the earlier the time, the smaller the side effects of the patient 's surgery on the patient.
postoperative pain score | One day after surgery
  The postoperative pain score of the patient was evaluated by the anesthesiologist. The postoperative pain score of the patient was evaluated by the postoperative anesthesia follow-up record in the medical record system. Minimum 0 points, maximum 100 points. The lower the score, the smaller the surgical trauma.
Postoperative patients were satisfied with the appearance | Two weeks after the operation
  The patient 's satisfaction with the operation was evaluated by the form of scale score. Minimum 0 points, maximum 100 points. The higher the score, the more satisfied the patient is with the operation.
The record of postoperative wound infection | Two weeks after the operation
  The record of postoperative wound infection is mainly recorded by the doctor during the postoperative follow-up. The occurrence of infection is a side effect of the operation.
The occurrence of postoperative wound fat liquefaction | Two weeks after the operation
  Postoperative wound fat liquefaction was mainly recorded by the doctor during postoperative follow-up. The occurrence of wound fat liquefaction was a side effect of surgery.
Postoperative wound peripheral nerve vascular injury | Two weeks after the operation
  The records of postoperative nerve injury were mainly recorded by doctors during postoperative follow-up. The occurrence of nerve injury is a side effect of surgery.
Postoperative incision hematoma formation | Two weeks after the operation
  The record of incision hematoma formation after operation is mainly recorded by doctors during postoperative follow-up. The occurrence of incision hematoma formation is a side effect of operation.

OTHER OUTCOMES:
Gluteal muscle contracture severity ZHAO 's classification | one day before surgery
  The ZHAO 's grading is evaluated by the physician according to the ZHAO 's grading scale. The lowest level of the scale is grade 1, and the highest level is grade 3. The higher the level, the more serious the gluteal muscle contracture is.
Demographic characteristics of patients | one day before surgery
  Demographic characteristics of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, the Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Considering the protection of patient privacy, we do not consider the disclosure of research data.

REFERENCES:
- [Result] Liu GH, Cao FQ, Yang SH, Zhu JF. Factors influencing the treatment of severe gluteal muscle contracture in children. J Pediatr Orthop B. 2011 Mar;20(2):67-9. doi: 10.1097/BPB.0b013e328341bcb2. PMID 21127436